CLINICAL TRIAL: NCT02591225
Title: Phenprocoumon Versus Dabigatran in Subjects With Atrial Fibrillation and Left Atrial Thrombus - a Prospective, Randomized, Controlled, Open-label One Year Follow-up Pilot Study
Brief Title: Left Atrial Thrombus Reduction - Effect of Dabigatran Versus Phenprocoumon
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Peter Bernhardt, Professor Dr., University of Ulm
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BI 1160.206
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Atrial Fibrillation; Left Atrial Thrombosis
Keywords: left atrial thrombus size; transesophageale echocardiography; silent cerebral embolism
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; Phenprocoumon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dabigatranetexilate (Experimental): Dabigatran capsula 150 mg; oral; bid; treatment period 12 months
  Interventions: Drug: Dabigatranetexilate
- Phenprocoumon (Active Comparator): Phenprocoumon INR adjusted; oral; once daily; treatment period 12 months
  Interventions: Drug: Phenprocoumon

INTERVENTIONS:
Drug: Dabigatranetexilate — After inclusion of the subjects with LA thrombus, they are treated according to the randomization either with Dabigatran (150 mg bid) or Phenprocoumon (INR adjusted once) for the treatment period of 12 months.
  Other Names: Pradaxa
  Arms: Dabigatranetexilate
Drug: Phenprocoumon — After inclusion of the subjects with LA thrombus, they are treated according to the randomization either with Dabigatran (150 mg bid) or Phenprocoumon (INR adjusted once) for the treatment period of 12 months.
  Other Names: Marcumar
  Arms: Phenprocoumon

SUMMARY:
This is a single-center, randomized, two treatment groups, open, phase IV clinical study in subjects with atrial fibrillation and left atrial thrombus. At Visit 0 (Screening Visit) subjects with left atrial thrombus established in transesophageal echocardiography (TEE) are eligible to entry in the study. If the subjects fulfill all other in- and exclusion criteria and undersign the informed consent the baseline cranial magnet resonance imaging (MRI) can be performed followed by randomization to one of the two treatment groups (Phenprocoumon or Dabigatran) at Visit 1 (Baseline Visit). The subjects will be treated for 12 months with Phenprocoumon (INR adjusted once daily) or Dabigatran 150 mg twice daily. Routinely clinical follow up visits will be done at week 4, month 3, month 6, month 9 and month 12. Follow up TEE will be performed after 4 weeks and after 12 months also the follow up cranial MRI at this visit. If the subject was randomized in the VKA group routinely INR measurements will performed.

DETAILED DESCRIPTION:
Bakground and study rationale: Left atrial (LA) thrombi are found in 2.5 - 18% of subjects with atrial fibrillation (AF) depending on the subject population. Subjects with LA thrombi have a particularly increased risk for cerebral and peripheral embolism. Consequently, oral anticoagulation is recommended in those subjects. Transesophageal echocardiography (TEE) is suited and is capable of visualizing and deecting LA thrombi. Cranial magnetic resonance imaging (MRI) has a high accurancy for detecting ailent cerebral mircoembolism. However, under continued effective anticoagulation with the vitamin K antagonist (VKA) Phenprocoumon we have shown that only 56% of LA thrombi resolve during a 12 months TEE observational period. At 1 month only 16% of the thrombi disappeared. However, cureent treatment guidelines recommend 4 weeks of effective anticoagulations prior cardioversion, independent of LA thrombus. In our subject population 84% of LA thrombi would have still been presented at 4 weeks VKA therapy and thus, would have had an increased risk of thromboembolism, if cardioversion, in accordance with current guidelines, would have performed. It is well known that thrombin plays a central role in the formation, growth, maintenance, and consolidation of thrombus. Direct thrombin inhibition has been shown to block these processes and leads to inhibition of thrombus. In vivo, it has been shown to reduce 90% of the preformed, half-hour-old-thrombus. This effect is probably due to better inhibition of the catalytically active clot-bound thrombin. Newer oral anticoagulants, like the direct thrombin inhibitor Dabigatran are therefore very promising for resolution of LA thrombi in comparison to VKA, which has not been investigated previously.

Efficacy variables: Expliration of possible differences for the reduction of left atrial thrombus size evaluated by TEE (primary) and silent cerebral embolism (secondary) detected by cranial MRI at baseline anf after a 12 month treated period with Phenprocoumon or Dabigatran in order to gain mire detailed information and to generate valid hypotheses for further clinical trials.

Overview: This is a single-center, randomized, two treatment groups, open, phase IV clinical study in subjects with atrial fibrillation and left atrial thrombus. At visit 0 (Screening visit) subjects with left atrial thrombus established in TEE are eligable to entry in the study. If the subjects fulfill all other in- and exclusion criteria and undersign the informed consent the baseline cranial MRI can be performed follwoed by randomization to one of the two treatment groups (Phenprocoumon or Dabigatran) at Visit 1 (Baseline visit). The subjects will be treated for 12 months with Phenprocoumon (INR adjusted once daily) or Dabigatran 150 mg twice daily. Routinly clinical follow up visits bill be done at week 4, month 3, month 6, month 9 and month 12. Follow up TEE will be performed after week 4 and month 12 also the follow up cranial MRI at this visit. If the subject was randomized in the VKA group routinely INR measurements will performed.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated written informed consent
* atrail fibrillation
* left atrial thrombus
* negative pregnancy test in woman with childbearin potentail
* subjects who have the ability to understand and comply the instructions for participation

Exclusion Criteria:

* low body weight < 50 kg
* instable cardiac or respiratory condition
* contraindication for Phenprocoumon or Dabigatran
* severely reduced renal function (CrCl < 30 ml/min)
* inadequate hepatic function (AST and ALT higher than 2 x ULN)
* Contraindication for MRI
* Durg/alcohol abusus
* Pregnant or nursing woman
* subject is an employee of any involved study investigator
* Parallel participation in another clinical trial
* Treatment with another investigational product

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
left atrial thrombus resolution | 12 months
  thrombus size evaluated by transeshophageal echocardiography

SECONDARY OUTCOMES:
cerebral emolism | 12 months
  cerebral embolic events detected by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bernhardt, MD, Principal Investigator — University Hospital Ulm, Department of Internal Medicine II
Locations (1):
- Department of Internal Medicine II, University Hospital Ulm, Ulm, Germany